CLINICAL TRIAL: NCT07193199
Title: A Novel Substrate and Injection Technique for Chin Augmentation
Brief Title: New Technique and Product for Chin Enhancement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-2025-RS
Record Dates: First submitted 2025-07-11; First posted 2025-09-25 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Aesthetic
Keywords: Hyaluronic Acid; Fillers; Facial Assessment; Chin Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Revanesse Sculpt+ (Other): Twenty-one (n = 21) male and female participants aged 18 years or older, including seven (n = 7) participants within each of the Allergan Chin Retrusion Scale(ACRS) categories corresponding to mild, moderate, and severe, based on the assessment of the Treating Investigator, will receive Revanesse Sculpt+ for the treatment of mild to severe chin retrusion at the Baseline visit (Visit 2) and will be eligible for retreatment 2 weeks later if a touch up is deemed necessary by the Treating Investigator. Volumes used for each participant will be determined by the aesthetic judgement of the Treating Investigator.
  Interventions: Device: Revanesse Sculpt+

INTERVENTIONS:
Device: Revanesse Sculpt+ — Revanesse Sculpt+ is approved and commercially available for use in Canada and is manufactured by Prollenium Technologies Inc. All study participants will receive Revanesse Sculpt+ for the treatment of mild to severe chin retrusion.

SUMMARY:
The use of hyaluronic acid (HA) fillers for soft tissue augmentation offers a valuable treatment modality for the correction of chin retrusion (i.e., when the chin appears to be set back or further back than normal in relation to the rest of the face). Their use is well-tolerated and provides satisfactory aesthetic results by improving facial balance and projection. Although the efficacy of hyaluronic acid HA fillers for chin augmentation has been established, the specific anatomy of the region may lead to adverse events. More specifically, certain fillers with strong integration characteristics may lead to product migration, while others with poor integration characteristics may lead to palpable deformities and distortion of the surrounding injection tissues.

Using a filler that has a high concentration of hyaluronic acid, a medium level of firmness and low water absorption may offer an effective option for treating this indication while minimizing certain adverse events. In addition, using consistent, standardized injection techniques can help achieve an ideal result.

We believe that the use of a novel HA gel (Revanesse Sculp+) for the chin, with a high concentration of HA, a moderate firmness and low water absorption, will perform better than historical controls with firmer properties in the management of chin retrusion.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, male and female participants 18 years of age and older;
2. Participants with established chin retrusion at Baseline (a score of minimal, moderate or severe; based on the Treating Investigator's Allergan Chin Retrusion Scale(ACRS)1 assessment;
3. Accepted the obligation not to receive any other facial procedures throughout the study duration;
4. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits;
5. No previous lower face fillers for 12 months prior to this study;
6. Capable of providing informed consent;
7. Willing to undergo scheduled CT scans as part of the study design;
8. Females of childbearing potential agree to take a scheduled urinary pregnancy test (UPT) prior to treatment administration.

Exclusion Criteria:

1. Participants without chin retrusion at Screening, per the ACRS1 ;
2. Participants with extreme chin retrusion at Screening as per the ACRS1;
3. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)];
4. Hypersensitivity to Revanesse products, hyaluronic acid filler or amide local anesthetics;
5. Participants presenting with porphyria or any other liver diseases;
6. Inability to comply with follow-up and abstain from facial injections during the study period;
7. Heavy smokers, classified as smoking more than 12 cigarettes per day;
8. History of severe or multiple allergies manifested by anaphylaxis, since drug allergies might preclude optimal management of complications;
9. Previous tissue revitalization therapy in the treatment area (i.e., the lower face) within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
10. Previous facial surgery, including liposuction;
11. Lifetime history of permanent implants in the treatment region (i.e., the lower face) including but not limited to dental implants;
12. Lifetime history of semi-permanent dermal fillers in the treatment region (i.e., the lower face);
13. History or presence of any disease or lesion near or at the treatment area, including inflammation, active or chronic infection, including in the mouth, dentals, head and neck region;
14. Active facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes zoster or any other facial condition that may increase the risk of cutaneous penetration of infective agents;
15. Scars, deformities, piercing, or tattoos in the treatment areas;
16. Facial cancer or precancer (e.g., actinic keratosis);
17. History of radiation therapy to the treatment area;
18. History of bleeding disorders, or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g., Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment;
19. Participants with immune disorders such as systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, and Hashimoto's thyroiditis, or participants using immunosuppressants;
20. Participants with a tendency to form hypertrophic or keloid scars, or any other healing disorders;
21. Participants with a tendency to form post-inflammatory hyperpigmentation;
22. Participants with known hypersensitivity to lidocaine or agents structurally related to amide type local anaesthetics (e.g., certain anti-arrhythmic);
23. Participants administered dental block or topical administration of lidocaine within 2 weeks of treatment;
24. Participants with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction;
25. Current remote infections (e.g., urinary tract, sinuses, intestinal tract, oral cavity);
26. Planned dental procedures during the 2-week period before and after filler treatments, including teeth cleaning, tooth extraction and gum grafts;
27. Planned vaccinations during the 2-week period before and after filler treatments;
28. Lifetime history of cystic acne, due to increased risk of cyst development following filler treatment;
29. CT scan reveals any bone-related abnormality (e.g., Osteoporosis, Paget's disease, bone infection or cancer), deformity, growths or anything in the Primary Investigator's opinion would interfere with the assessment of any endpoint;
30. Participant is undergoing orthodontic procedures/treatments that manipulate the teeth and underlying bone structure including but not limited to braces and Invisalign treatments;
31. Participants who cannot/should not, for any reason (medical or otherwise), undergo scheduled CT scans (i.e., due to increased safety risks);
32. History of clinically significant medical conditions or any other reason that the investigator determines would interfere with the participants participation in this study or would make the participant an unsuitable candidate to receive study medical device;

    * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
    * History of facial nerve palsy
    * Infection or dermatological condition at the treatment injection sites
    * Marked facial dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or excessively photodamaged skin
33. Participant has an anticipated need for overnight hospitalization or scheduled surgery;
34. Participant has been treated with any other investigational product at least 30 days before the first administration of the current investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Frequency of participants graded as at least 'improved' on the Global Aesthetic Improvement Scale (GAIS) by a blinded evaluator at baseline to Month 12 | Baseline to Month 12
  Frequency of participants having at least "improved" (e.g., "improved", "much improved" or "very much improved") on the Global Aesthetics Improvement Scale (GAIS), as graded by a blinded evaluator.
  The Global Aesthetics Improvement Scale (GAIS) is a five-point Likert scale, categorized as "worse", "no change", "improved", "much improved" and "very much improved".
Proportion of participants with ≥1 grade-point improvement from baseline in chin retrusion, as assessed by a blinded evaluator using the CCPS and/or ACRS | Baseline to Month 12
  The Croma Chin Projection Assessment Scale (CCPS) is a a validated 5-point assessment tool for the projection of the chin using a vertical line from pogonium through the lower vermilion boarder in front of the labiomental crease. It grades chin retrusion from 0 (ideal chin projection) to 4 (very severe retrusion).
  The Allergan Chin Retrusion Scale (ACRS) is a validated 5-point assessment tool for chin retrusion using the midpoint of the chin and the lower vermillion boarder. It grades chin retrusion from 0 (no retrusion) to 4 (extreme chin retrusion).

SECONDARY OUTCOMES:
Frequency of post-injection reactions including pain and discomfort during treatment, immediately after treatment, and at 14 days post-treatment | Baseline to Month 12
  Frequency of post injection reactions including pain and discomfort (generalized, during chewing, talking, and/or kissing as applicable) during treatment, immediately after treatment and 14 days following treatment.
Frequency of physician-reported and participant-reported adverse events (AEs) at any visit post-injection | Baseline to Month 12
  Frequency of post injections reactions including physician-reported and participant-reported adverse events (AEs) at any visit.

OTHER OUTCOMES:
Change perimental tissue depth assessed by CT imaging at Months 6 and 12 compared to baseline | Baseline, Month 6, Month 12
  The degree of changes in peri-injection tissue will be observed through computed tomography (CT) scans at Months 6 and 12, compared to Baseline, and will be evaluated by a blinded radiologist using a depth quantification (mm) assessment.
Correlation between hyaluronic acid (HA) volume injected and the incidence and/or severity of HA-related tissue changes in the chin at Months 6 and 12 | Baseline, Month 6, Month 12
  The correlation between HA volumes used and the incidence and/or severity of HA-related tissue changes in the chin area observed through computed tomography (CT) scans at Months 6 and 12, compared to Baseline, will be analyzed.
Correlation between aesthetic improvement and degree of tissue changes in the chin area from Baseline to Month 12 | Baseline to Month 12
  Correlation between depth of chin tissue changes (mm), and change in aesthetic outcomes, as measured by at least 1 grade point decrease in the Global Aesthetic Improvement Scale (GAIS) at any visit, will be analyzed.
Proportion of Participants Reporting being at least satisfied with treatment after Treatment using a 7-point Likert Scale from Week 2 to Month 12 | Week 2 to Month 12
  Change in participant satisfaction with treatment will be evaluated using a 7-point Likert scale (extremely satisfied, very much satisfied, satisfied, neutral, dissatisfied, very much dissatisfied, extremely dissatisfied) at study visits Week 2 to Month 12.
Change in participant satisfaction of their chin using the FACE-Q questionnaire as assessed from baseline to Month 12 | Baseline to Month 12
  The FACE-Q Satisfaction with Chin questionnaire will be used to evaluate participant satisfaction with their chin at all visits from Baseline to Month 12.
Change in participant satisfaction with facial balance (facial thirds) as assessed using a 5-point Likert scale form from Baseline to Month 12 | Baseline to Month 12
  The participant satisfaction with facial balance and changes to the facial thirds (upper, middle, lower face) will be evaluated at all visits using a five-point Likert scale (very much satisfied, satisfied, neutral, unsatisfied, very much unsatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, PhD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No